CLINICAL TRIAL: NCT00916526
Title: Measurement of Exhaled NO and Bronchial Provocation Test With Mannitol as a Predictor of Response to Inhaled Corticosteroids in Chronic Cough
Brief Title: Measurement of Exhaled Nitric Oxide (NO) and Bronchial Provocation Test With Mannitol as a Predictor of Response to Inhaled Corticosteroids in Chronic Cough
Acronym: MANOTOUX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Syntara (Industry)
Responsible Party: Clément Caillaux, CHU de Saint-Etienne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0808078; 2008-A00846-49 (Other: AFSSAPS)
Record Dates: First submitted 2009-06-08; First posted 2009-06-09 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Cough; Bronchial Hyperreactivity
Keywords: Chronic cough; Inhaled corticosteroid treatment; Bronchial provocation test with mannitol; Methacholine
MeSH Terms: conditions — Cough; Bronchial Hyperreactivity; Chronic Cough | interventions — Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bronchial provocation test with mannitol (Experimental): Patients referred for evaluation of a chronic cough (without treatment or after stopping inhaled corticosteroids for 2 weeks) will perform a measure of FeNO, a bronchial provocation test with mannitol, will fill out a questionnaire of quality of life for the cough (Leicester Cough Questionnaire) and the intensity of coughing on a 10-cm visual scale.
  After 6 weeks after treatment with inhaled corticosteroids patients will perform the same tests.
  Interventions: Procedure: bronchial provocation test with mannitol

INTERVENTIONS:
Procedure: bronchial provocation test with mannitol — Bronchial provocation test with mannitol: Aridol is supplied in kit form containing sufficient capsules to complete one complete challenge, and the inhalation device.
  1. Apply nose clip and subject should be directed to breathe through the mouth
  2. Insert 0 mg capsule into inhalation device. Puncture capsule by depressing buttons on side of device slowly, and once only (a second puncture may fragment the capsules)
  3. The patient should exhale completely, before inhaling from device in a controlled rapid deep inspiration
  4. At the end of deep inspiration, start 60 second timer, subject should hold breath for 5 seconds and exhale through mouth before removal of nose clip
  5. At the end of 60 seconds, measure the FEV1 in duplicate (this becomes baseline FEV1)
  6. Insert 5 mg capsule into inhalation device, and proceed as above
  7. Repeat steps 1 - 4 following the dose steps in the table below until the patient has a positive response or 635 mg has been administered.
  Other Names: Aridol

SUMMARY:
Chronic cough is defined by its persistence beyond 8 weeks. Many conditions can explain the existence of a bronchial inflammation. In the management of chronic cough, the search for bronchial hyperreactivity (HRB) is recommended. The treatment relies primarily on the prescription of inhaled corticosteroids. It has been shown recently that the existence of an HRB with Methacholine (bronchial provocation test used in routine) does predict the effectiveness of inhaled corticosteroid treatment in no more than 50% of cases.

It is now possible to assess the bronchial inflammation by rapid, non-invasive and reproducible tests such that the fraction of exhaled nitric oxide (FeNO) and bronchial provocation test with mannitol. In a retrospective study, it was shown that an increased value of FeNO (cut-off > 35 ppb) predicts a positive response to treatment with a sensitivity of 90% and a specificity of 80%.

DETAILED DESCRIPTION:
The purpose of this study is to show that the use of the prospective value of exhaled NO can predict response to treatment with inhaled corticosteroids in adult with chronic cough. In addition we will assess the interest of the prognosis of bronchial provocation test with mannitol in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Cough during 2 months
* Social Security regimen affiliated
* Consent form signed

Exclusion Criteria:

* Smoking active
* Treatment with angiotensin converting enzyme inhibitor
* Clinical signs of obvious gastroesophageal reflux
* Clinical rhinosinusitis
* Recent respiratory infection (< 1 month)
* Corticosteroid Treatment(oral or inhaled) within 2 weeks
* VEMS < 1 L or < 80% of the theoretical value
* Existence of an obstructive ventilatory disorder defined as a report (FEV/FVC) < 90% of the theoretical value

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The intensity of coughing on a 10-cm visual scale | 6 weeks after treatment with inhaled corticosteroids

SECONDARY OUTCOMES:
Sensitivity, specificity, positive predictive value and negative predictive value of the threshold value of 35 ppb FeNo to the clinical response seen as positive if the EVA reduces cough of at least 2 cm | 6 weeks after treatment with inhaled corticosteroids
Sensitivity, specificity, positive predictive value and negative predictive value of response to bronchial provocation test with mannitol on the clinical response seen as positive if the EVA reduces cough of at least 2 cm | 6 weeks after treatment with inhaled corticosteroids
Correlation between the value of FeNo and dose of mannitol causing a fall of 15% of maximum volume expired second (PD15) | 6 weeks after treatment with inhaled corticosteroids
Score quality of life of the Leicester Cough Questionnaire | 6 weeks after treatment with inhaled corticosteroids

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric COSTES, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France